## The Effect of Word Characteristics and Orthography on Vocabulary Learning NCT # Not yet assigned

Version of document completed 1

Statistical Analysis Plan

## **Statistical Analyses**

The most recent Statistical Packages for the Social Sciences (SPSS) version 28 will be used to perform separate repeated-measures analyses of covariance (ANCOVA) to explore the main effects and interactions between phonotactic probability (PP; high/low) and orthography (present/absent) on vocabulary comprehension, recognition, production, spelling recognition, and spelling production. Mother's years of education served as the covariate when included.

## **Levels and Factors**

Levels refer to the different categories or conditions within a factor. Each factor can have two or more levels. This study involves two key factors: PP and orthography. Each factor is characterized by two distinct levels. For PP, the levels are defined as high versus low, reflecting the probability of a particular phonotactic pattern occurring within words. For orthography, the levels are defined as the presence or absence of orthography.

## **Dependent Variables**

Research Question 1 - Is there a significant difference in total correct scores at post-test for different word types with or without orthography with pre-test scores and mother's education level covaried as measured by comprehension, recognition, production, spelling recognition, and spelling production?

A repeated measures ANOVA was conducted. The between-subjects factor is PP and Orthography. the word type (1 = high with orth; 2 = highwithout; 3 =lowwith; 4= lowwithout). The within subjects variable is total correct scores in the pretest and post test. The covariate is mothers educational level.